CLINICAL TRIAL: NCT02919306
Title: A Combined Phase 1/2a, Exploratory Study of a Therapeutic Vaccine Using an Adenovirus Type 26 Vector Prime and Modified Vaccinia Ankara Boost Combination With Mosaic Inserts in HIV-1 Infected Adults Who Initiated Antiretroviral Treatment During Acute HIV Infection
Brief Title: Safety and Efficacy Study of Vaccine Schedule With Ad26.Mos.HIV and MVA-Mosaic in Human Immunodeficiency Virus (HIV)-Infected Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108161; VAC89220HTX1001 (Other: Janssen Vaccines & Prevention B.V.)
Record Dates: First submitted 2016-09-01; First posted 2016-09-29 (Estimated); Results first posted 2022-03-11 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Ad26.Mos.HIV Vaccine or MVA mosaic Vaccine (Experimental): Participants will receive adenovirus serotype 26-Mosaic -Human Immunodeficiency Virus (Ad26.Mos.HIV) 0.5 milliliter (mL) injection intramuscularly (containing 5 * 10^10 viral particles [vp]) at Weeks 0 and 12 followed by modified Vaccinia Ankara-Mosaic (MVA mosaic) 0.5 mL injection (containing 10^8 Plaque-forming unit [pfu]) at Week 24 and 48.
  Interventions: Biological: Ad26.Mos.HIV; Biological: MVA-Mosaic
- Placebo (Placebo Comparator): 0.5 mL Sodium Chloride Injection United States Pharmacopeia (USP) 0.9% will be administered by intramuscular (IM) injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Ad26.Mos.HIV — Recombinant replication-deficient Ad26 vectored vaccine and consists of 3 Ad26 vectors, one containing a mosaic insert of envelope (Env) sequence, and 2 vectors containing mosaic inserts of Gag and Pol sequences (Ad26.Mos.1.Env + Ad26.Mos1.Gag-Pol + Ad26.Mos2.Gag-Pol). Total dose is 5*10^10 viral particle per 0.5 milliliter (mL) injection administered intramuscularly.
  Arms: Ad26.Mos.HIV Vaccine or MVA mosaic Vaccine
Biological: MVA-Mosaic — Recombinant live attenuated MVA virus-vectored vaccine that has been genetically engineered to express 2 mosaic Gag, Pol, and Env sequences (Mosaic 1 and Mosaic 2). Total dose is 10^8 plaque-forming unit per 0.5 mL injection administered intramuscularly.
  Arms: Ad26.Mos.HIV Vaccine or MVA mosaic Vaccine
Drug: Placebo — Participants will receive placebo intramuscularly Weeks 0, 12, 24 and 48.
  Arms: Placebo

SUMMARY:
The purpose of the study is to assess: 1 safety and tolerability of adenovirus serotype 26 (Ad26) prime and Modified Vaccinia Ankara (MVA) boost versus placebo in participants on suppressive antiretroviral therapy (ART) that was initiated during acute Human Immunodeficiency Virus (HIV) infection; 2) Measure the frequency and duration of sustained viremic control after receiving Ad26 prime/MVA boost or placebo, defined as greater than 24 weeks with plasma HIV ribonucleic acid (RNA) lesser than (<)50 copies/ml after antiretroviral (ARV) analytical treatment interruption (ATI).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed human immunodeficiency virus (HIV)-1 infected and started antiretroviral therapy (ART) during acute infection (Fiebig stages I, II, III or IV) as part of trial RV254
* Treatment with current stable antiretroviral therapy (ART) (no changes to treatment) for at least 4 weeks prior to screening
* All female participants of childbearing potential must have a negative serum pregnancy test (beta human chorionic gonadotropin) at the screening visit, and a negative urine pregnancy test prior to vaccination on Day 1 and prior to subsequent study vaccinations
* HIV ribonucleic acid (RNA) less than (<)50 copies per milliliter (copies/ml) for at least 48 weeks at screening: a) One blip of HIV RNA greater than (>)50 and <200 copies/ml within 48 weeks is acceptable, provided that the most recent (before screening) HIV RNA <50 copies/ml
* Laboratory criteria during screening: a) Hemoglobin: Women: greater than or equal to >=11 gram/deciliter (g/dL); Men >=12.5 g/dL, b) White cell count: 2,500 to 11,000 cells per cubic millimeter (cells/mm^3), c) Platelets: 125,000 to 450,000 per mm^3, d) Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less than or equal to <=1.5x institutional upper limits of normal (ULN), e) Creatinine <=1.5x institutional ULN, f) CD4 > 400 cells/mm^3, g) Troponin <1x ULN
* A woman must be either: a) Not of childbearing potential: postmenopausal (>45 years of age with amenorrhea for at least 2 years, or any age with amenorrhea for at least 6 months and a serum follicle stimulation hormone [FSH] level >40 International Units Per Liter (IU/L); surgically sterile; or b) Of child-bearing potential and practicing an effective double method of birth control (example, prescription oral contraceptives, contraceptive injections, intrauterine device, contraceptive patch, or vaginal ring, in conjunction with either a female condom or one of the methods for male contraception before entry and through 3 months after the last vaccination

Exclusion Criteria:

* Receipt of any vaccine within 30 days prior to the first vaccination or plans to receive within 30 days post-vaccination. In the case of medically indicated vaccines, the vaccination should be given at least 2 weeks before or after the first vaccination. However, if a vaccine is indicated in a post exposure setting (example, rabies or tetanus), it must take priority over the study vaccine and same rules will apply to subsequent study vaccinations
* Any history of HIV-related illness under Centers for Disease Control and Prevention (CDC) category C
* History of myocarditis, pericarditis, cardiomyopathy, congestive heart failure with permanent sequelae, clinically significant arrhythmia (including any arrhythmia requiring medication, treatment, or clinical follow-up)
* Chronic active hepatitis B or active hepatitis C (for example, positive serology with confirmatory positive polymerase chain reaction) or active syphilis infection. Active syphilis documented by examination or serology unless positive serology is due to past treated infection
* Receipt of blood products or immunoglobulin in the past 3 months
* History of anaphylaxis or other serious adverse reactions to vaccines or vaccine products, or neomycin or streptomycin or egg products
* History of chronic urticaria (recurrent hives)
* Chronic or recurrent use of medications which modify host immune response, example (e.g.) cancer chemotherapeutic agents, parenteral corticosteroids (short course oral steroids given for non-chronic conditions not expected to recur is not an exclusion criteria, topical steroid use is not an exclusion criteria), etc. but not including ART

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (1):
- Bangkok, Thailand

REFERENCES:
- [Derived] Kroon E, Chottanapund S, Buranapraditkun S, Sacdalan C, Colby DJ, Chomchey N, Prueksakaew P, Pinyakorn S, Trichavaroj R, Vasan S, Manasnayakorn S, Reilly C, Helgeson E, Anderson J, David C, Zulk J, de Souza M, Tovanabutra S, Schuetz A, Robb ML, Douek DC, Phanuphak N, Haase A, Ananworanich J, Schacker TW. Paradoxically Greater Persistence of HIV RNA-Positive Cells in Lymphoid Tissue When ART Is Initiated in the Earliest Stage of Infection. J Infect Dis. 2022 Jun 15;225(12):2167-2175. doi: 10.1093/infdis/jiac089. PMID 35275599
- [Derived] Colby DJ, Sarnecki M, Barouch DH, Tipsuk S, Stieh DJ, Kroon E, Schuetz A, Intasan J, Sacdalan C, Pinyakorn S, Grandin P, Song H, Tovanabutra S, Shubin Z, Kim D, Paquin-Proulx D, Eller MA, Thomas R, de Souza M, Wieczorek L, Polonis VR, Pagliuzza A, Chomont N, Peter L, Nkolola JP, Vingerhoets J, Truyers C, Pau MG, Schuitemaker H, Phanuphak N, Michael N, Robb ML, Tomaka FL, Ananworanich J. Safety and immunogenicity of Ad26 and MVA vaccines in acutely treated HIV and effect on viral rebound after antiretroviral therapy interruption. Nat Med. 2020 Apr;26(4):498-501. doi: 10.1038/s41591-020-0774-y. Epub 2020 Mar 23. PMID 32235883
- See also: Manual upload due to format issue between PRS and PCM. — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR108161&attachmentIdentifier=1ee00b92-049e-4ea6-8b76-3014743e665b&fileName=CR108161_DownloadReceipt_Initial_Results.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 37 participants screened for this study, 27 participants were randomized and received at least 1 dose of active vaccine (18 participants) or placebo (9 participants). One participant in the active vaccine group was excluded from the analysis on request of the Ethics Committee due to a major protocol deviation.
Groups:
- Ad26.Mos.HIV Vaccine or MVA Mosaic Vaccine: Participants from study NCT03032575, NCT01397669, NCT02475915, NCT02750059, and NCT00796146 who started on antiretroviral therapy (ART) during acute human immunodeficiency virus (HIV) infection, and who were on a current stable ART for at least 4 weeks prior to screening received adenovirus serotype 26-Mosaic -Human Immunodeficiency Virus (Ad26.Mos.HIV) 0.5 milliliter (mL) injection intramuscularly (IM) (containing 5*10^10 viral particles [vp]) at Weeks 0 and 12 followed by modified Vaccinia Ankara-Mosaic (MVA mosaic) 0.5 mL injection (containing 10^8 Plaque-forming unit [pfu]) at Weeks 24 and 48 (Stage 1). Participants who met immunologic response criteria (more than 50 percent [%] of vaccines had an increase of Interferon [IFN]-gamma producing cells) (36 weeks of follow-up) were verified at Week 60 (Stage 2). For eligible participants, an analytical treatment interruption (ATI) was started and all ARTs were discontinued. Participants had to reinitiate ART after ATI using the same regimen as their previous treatment (before Week 60) when Human Immunodeficiency Virus-1 (HIV-1) Ribonucleic Acid (RNA) more than (>) 1,000 copies per milliliters (copies/mL) twice at least 1 week apart or cluster of differentiation (CD) 4+ T cell counts less than (<) 350 per cubic millimeter (350/mm^3) twice at least 2 weeks apart or CD4+ T cell count decline of > 50% from Week 60 prior to ATI up to Week 96.
- Placebo: Participants from study RV254 who started on ART during acute HIV infection, who were on a current stable ART for at least 4 weeks prior to screening received placebo IM injection at Weeks 0, 12, 24, and 48 (Stage 1). Participants who met immunologic response criteria (more than 50% vaccines had an increase of IFN-gamma producing cells in the vaccine arm) (36 weeks of follow-up) were verified at Week 60 (Stage 2). For eligible participants, an ATI was started and all ARTs were discontinued. Participants had to reinitiate ART after ATI using the same regimen as their previous treatment (before Week 60) when HIV-1 RNA >1,000 copies/mL twice at least 1 week apart or CD 4+ T cell counts <350/mm^3 twice at least 2 weeks apart or CD4+ T cell count decline of > 50% from Week 60 prior to ATI up to Week 96.
Period: Overall Study
Arm/Group | Ad26.Mos.HIV Vaccine or MVA Mosaic Vaccine | Placebo
Started | 18 | 9
Completed | 16 | 9
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ad26.Mos.HIV Vaccine or MVA Mosaic Vaccine | Placebo | Total
Number analyzed (Participants) | 17 | 9 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.4 (5.39) | 26.3 (6.87) | 27 (5.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 17 | 9 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 17 | 9 | 26
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  THAILAND | 17 | 9 | 26

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Grade 3 or 4 Solicited Local Adverse Events (AEs)
Description: Solicited local AE of grade 3 or 4 and that is thought to be related to study vaccine were reported. An AE is any untoward medical occurrence in a clinical study participant administered a investigational or non-investigational medicinal product. An AE does not necessarily have a causal relationship with the treatment. Solicited local AEs (at injection site) included pain/tenderness, erythema, induration, swelling, itching and warmth were collected and reported for 7 days after each vaccination.
Time Frame: Up to Week 49 (7 days post each vaccination)
Population: FAS included all participants who were randomized and who received at least 1 dose of study vaccine or placebo.
Measure: Number; unit: percentage of participants
Arm/Group | Ad26.Mos.HIV Vaccine or MVA Mosaic Vaccine | Placebo
Number analyzed (Participants) | 17 | 9
percentage of participants | 0 | 0

2. Primary Outcome: Percentage of Participants With Grade 3 or 4 Solicited Systemic AEs
Description: Solicited systemic AE of grade 3 or 4 and that is thought to be related to study vaccine were reported. Solicited systemic AEs included fever (defined as body temperature of 38.0-degree celsius or higher), fatigue, headache, myalgia, arthralgia, chills, nausea, vomiting, rashes, and general itching.
Time Frame: Up to Week 49 (7 days post each vaccination)
Population: FAS included all participants who were randomized and who received at least 1 dose of study vaccine or placebo.
Measure: Number; unit: percentage of participants
Arm/Group | Ad26.Mos.HIV Vaccine or MVA Mosaic Vaccine | Placebo
Number analyzed (Participants) | 17 | 9
percentage of participants | 0 | 0

3. Primary Outcome: Percentage of Participants With Grade 3 or 4 Unsolicited AEs
Description: Unsolicited AE with worst severity grade 3 or 4 and that is thought to be related to study vaccine were reported. Unsolicited AEs were defined as events that participants experienced but were not specifically asked about.
Time Frame: Up to Week 52 (28 days after each vaccination)
Population: FAS included all participants who were randomized and who received at least 1 dose of study vaccine or placebo.
Measure: Number; unit: percentage of participants
Arm/Group | Ad26.Mos.HIV Vaccine or MVA Mosaic Vaccine | Placebo
Number analyzed (Participants) | 17 | 9
percentage of participants | 0 | 0

4. Primary Outcome: Percentage of Participants With Grade 3 or 4 Related AEs
Description: Related AEs of grade 3 or 4 and that is thought to be related to study vaccine were reported.
Time Frame: Up to Week 52 (28 days after each vaccination)
Population: FAS included all participants who were randomized and who received at least 1 dose of study vaccine or placebo.
Measure: Number; unit: percentage of participants
Arm/Group | Ad26.Mos.HIV Vaccine or MVA Mosaic Vaccine | Placebo
Number analyzed (Participants) | 17 | 9
percentage of participants | 0 | 0

5. Primary Outcome: Percentage of Participants With Solicited Local AEs for 7 Days After Each Vaccination
Description: An AE is any untoward medical occurrence in a clinical study participant administered a investigational or non-investigational medicinal product. An AE does not necessarily have a causal relationship with the treatment. Solicited local AEs (at injection site) included pain/tenderness, erythema, induration, swelling, itching and warmth were collected and reported for 7 days after each vaccination.
Time Frame: Up to Week 49 (7 days post each vaccination)
Population: The Full Analysis Set (FAS) included all participants who were randomized and who received at least 1 dose of study vaccine or placebo.
Measure: Number; unit: percentage of participants
Arm/Group | Ad26.Mos.HIV Vaccine or MVA Mosaic Vaccine | Placebo
Number analyzed (Participants) | 17 | 9
percentage of participants | 88.2 | 66.7

6. Primary Outcome: Percentage of Participants With Solicited Systemic AEs for 7 Days After Each Vaccination
Description: Solicited systemic AEs included fever (defined as body temperature of 38.0-degree celsius or higher), fatigue, headache, myalgia, arthralgia, chills, nausea, vomiting, rashes, and general itching were collected and reported for 7 days after each vaccination.
Time Frame: Up to Week 49 (7 days after each vaccination)
Population: FAS included all participants who were randomized and who received at least 1 dose of study vaccine or placebo.
Measure: Number; unit: percentage of participants
Arm/Group | Ad26.Mos.HIV Vaccine or MVA Mosaic Vaccine | Placebo
Number analyzed (Participants) | 17 | 9
percentage of participants | 70.6 | 55.6

7. Primary Outcome: Percentage of Participants With Unsolicited AEs 28 Days After Each Vaccination
Description: Unsolicited AEs were defined as events that participants experienced but were not specifically asked about.
Time Frame: Up to Week 52 (28 days after each vaccination)
Population: FAS included all participants who were randomized and who received at least 1 dose of study vaccine or placebo.
Measure: Number; unit: percentage of participants
Arm/Group | Ad26.Mos.HIV Vaccine or MVA Mosaic Vaccine | Placebo
Number analyzed (Participants) | 17 | 9
percentage of participants | 88.2 | 77.8

8. Primary Outcome: Percentage of Participants With Related AEs and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant administered a investigational or non-investigational medicinal product. An AE does not necessarily have a causal relationship with the treatment. A SAE is any AE that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect and is a suspected transmission of any infectious agent via a medicinal product.
Time Frame: Up to Week 52 (28 days after each vaccination)
Population: FAS included all participants who were randomized and who received at least 1 dose of study vaccine or placebo.
Measure: Number; unit: percentage of participants
Arm/Group | Ad26.Mos.HIV Vaccine or MVA Mosaic Vaccine | Placebo
Number analyzed (Participants) | 17 | 9
percentage of participants
  Related AEs | 29.4 | 0
  Related SAEs | 0 | 0

9. Primary Outcome: Percentage of Participants With AEs Leading to Discontinuation of Study Vaccination
Description: Percentage of participants with AEs leading to discontinuation of study vaccination were reported.
Time Frame: Up to Week 96
Population: FAS included all participants who were randomized and who received at least 1 dose of study vaccine or placebo.
Measure: Number; unit: percentage of participants
Arm/Group | Ad26.Mos.HIV Vaccine or MVA Mosaic Vaccine | Placebo
Number analyzed (Participants) | 17 | 9
percentage of participants | 0 | 0

10. Primary Outcome: Percentage of Participants With AEs
Description: Percentage of participants with AEs were reported.
Time Frame: Up to Week 52 (28 days after each vaccination)
Population: FAS included all participants who were randomized and who received at least 1 dose of study vaccine or placebo. The data was planned for unsolicited AEs during the 28-day post-vaccination phase.
Measure: Number; unit: percentage of participants
Arm/Group | Ad26.Mos.HIV Vaccine or MVA Mosaic Vaccine | Placebo
Number analyzed (Participants) | 17 | 9
percentage of participants | 88.2 | 77.8

11. Primary Outcome: Percentage of Participants With Worst Laboratory Toxicity Grades 1, 2, 3, and 4 and Non-graded Serum Chemistry Abnormalities
Description: Percentage of participants with worst laboratory grades 1 (mild), 2 (moderate), 3 (severe), and 4 (potentially life-threatening) and non-graded serum chemistry abnormalities were reported. Serum chemistry parameters included alanine aminotransferase, aspartate aminotransferase, creatine, hyperglycemia, hypoglycemia, gamma-gutamyl transferase, chloride, urea nitrogen, and bilirubin. The parameters not represented in the grading scale, abnormalities were indicated as being 'high' or 'low' or 'abnormal'.
Time Frame: Up to Week 96
Population: FAS included all participants who were randomized and who received at least 1 dose of study vaccine or placebo. Here 'n' (number analyzed) signifies number of participants evaluable for specified categories.
Measure: Number; unit: percentage of participants
Arm/Group | Ad26.Mos.HIV Vaccine or MVA Mosaic Vaccine | Placebo
Number analyzed (Participants) | 17 | 9
percentage of participants
  Post-Any Dose: Alanine Aminotransferase- Grade 1: number analyzed (Participants) | 2 | 0
  Post-Any Dose: Alanine Aminotransferase- Grade 1 | 50 |
  Post-Any Dose: Alanine Aminotransferase- Grade 3: number analyzed (Participants) | 2 | 0
  Post-Any Dose: Alanine Aminotransferase- Grade 3 | 50 |
  Post-Any Dose: Aspartate Aminotransferase- Grade 1: number analyzed (Participants) | 2 | 0
  Post-Any Dose: Aspartate Aminotransferase- Grade 1 | 50 |
  Post-Any Dose: Aspartate Aminotransferase- Grade 4: number analyzed (Participants) | 2 | 0
  Post-Any Dose: Aspartate Aminotransferase- Grade 4 | 50 |
  ART resumption: Alanine Aminotransferase- Grade 1: number analyzed (Participants) | 16 | 8
  ART resumption: Alanine Aminotransferase- Grade 1 | 12.5 | 12.5
  ART resumption: Aspartate Aminotransferase- Grade 1: number analyzed (Participants) | 16 | 8
  ART resumption: Aspartate Aminotransferase- Grade 1 | 12.5 | 37.5
  ART resumption: Creatine- Grade 1: number analyzed (Participants) | 16 | 8
  ART resumption: Creatine- Grade 1 | 12.5 | 25
  ART resumption: Hyperglycemia- Grade 1: number analyzed (Participants) | 16 | 8
  ART resumption: Hyperglycemia- Grade 1 | 6.3 | 0
  ART resumption: Hyperglycemia- Grade 2: number analyzed (Participants) | 16 | 8
  ART resumption: Hyperglycemia- Grade 2 | 6.3 | 0
  ART resumption: Hypoglycemia- Grade 1: number analyzed (Participants) | 16 | 8
  ART resumption: Hypoglycemia- Grade 1 | 0 | 12.5
  ART resumption: Hypoglycemia- Grade 2: number analyzed (Participants) | 16 | 8
  ART resumption: Hypoglycemia- Grade 2 | 6.3 | 0
  ATP: Gamma Glutamyl Transferase (high) | 5.9 | 11.1
  ATP: Gamma Glutamyl Transferase (low) | 0 | 11.1
  ART resumption: Chloride (High) | 18.8 | 12.5
  ART resumption: Gamma Glutamyl Transferase (Low) | 6.3 | 0
  ART resumption: Urea Nitrogen (Low): number analyzed (Participants) | 16 | 8
  ART resumption: Urea Nitrogen (Low) | 12.5 | 0
  ART Resumption: Bilirubin: number analyzed (Participants) | 16 | 8
  ART Resumption: Bilirubin | 0 | 12.5

12. Primary Outcome: Percentage of Participants With Worst Laboratory Toxicity Grade 1 and Non-graded Hematology Abnormalities
Description: Percentage of participants with worst laboratory toxicity grade 1 (mild) and non-graded hematology abnormalities were reported. Hematology parameters included absolute neutrophil count, basophils/leukocytes, eosinophils/leukocytes, hematocrit, lymphocytes/leukocytes, monocytes/leukocytes, neutrophils/leukocytes, erythrocytes, hematocrit, neutrophils, basophils, eosinophils, eosinophils/leukocytes, monocytes, neutrophils and platelet count. The parameters not represented in the grading scale, abnormalities were indicated as being 'high' or 'low' or 'abnormal'.
Time Frame: Up to Week 96
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Ad26.Mos.HIV Vaccine or MVA Mosaic Vaccine | Placebo
Number analyzed (Participants) | 17 | 9
percentage of participants
  ART resumption: Absolute Neutrophil Count-Grade 1: number analyzed (Participants) | 17 | 8
  ART resumption: Absolute Neutrophil Count-Grade 1 | 0 | 12.5
  Post-Any Dose: Basophils/Leukocytes (high) | 11.8 | 0
  Post-Any Dose: Eosinophils/Leukocytes (high) | 5.9 | 11.1
  Post-Any Dose: Hematocrit (low) | 5.9 | 11.1
  Post-Any Dose: Lymphocytes/Leukocytes (high) | 0 | 11.1
  Post-Any Dose: Lymphocytes/Leukocytes (low) | 5.9 | 0
  Post-Any Dose: Monocytes/Leukocytes (high) | 5.9 | 11.1
  Post-Any Dose: Neutrophils/Leukocytes (low) | 5.9 | 11.1
  ATI: Eosinophils/Leukocytes (high) | 0 | 33.3
  ATI: Eosinophils/Leukocytes (low) | 0 | 11.1
  ATI: Erythrocytes (low) | 17.6 | 11.1
  ATI: Hematocrit (low) | 23.5 | 11.1
  ATI: Lymphocytes/Leukocytes (high) | 5.9 | 22.2
  ATI: Lymphocytes/Leukocytes (low) | 0 | 11.1
  ATI: Monocytes/Leukocytes (high) | 35.3 | 44.4
  ATI: Neutrophils (low) | 11.8 | 11.1
  ATI: Neutrophils/Leukocytes (low) | 5.9 | 22.2
  ART resumption: Basophils (high): number analyzed (Participants) | 17 | 8
  ART resumption: Basophils (high) | 0 | 12.5
  ART resumption: Basophils/Leukocytes (high): number analyzed (Participants) | 17 | 8
  ART resumption: Basophils/Leukocytes (high) | 11.8 | 25
  ART resumption: Eosinophils (high): number analyzed (Participants) | 17 | 8
  ART resumption: Eosinophils (high) | 0 | 12.5
  ART resumption: Eosinophils (low): number analyzed (Participants) | 17 | 8
  ART resumption: Eosinophils (low) | 17.6 | 12.5
  ART resumption: Eosinophils/Leukocytes (high): number analyzed (Participants) | 17 | 8
  ART resumption: Eosinophils/Leukocytes (high) | 11.8 | 37.5
  ART resumption: Eosinophils/Leukocytes (low): number analyzed (Participants) | 17 | 8
  ART resumption: Eosinophils/Leukocytes (low) | 17.6 | 12.5
  ART resumption: Erythrocytes (high): number analyzed (Participants) | 17 | 8
  ART resumption: Erythrocytes (high) | 5.9 | 0
  ART resumption: Erythrocytes (low): number analyzed (Participants) | 17 | 8
  ART resumption: Erythrocytes (low) | 11.8 | 12.5
  ART resumption: Hematocrit (low): number analyzed (Participants) | 17 | 8
  ART resumption: Hematocrit (low) | 29.4 | 12.5
  ART resumption: Lymphocytes/Leukocytes (high): number analyzed (Participants) | 17 | 8
  ART resumption: Lymphocytes/Leukocytes (high) | 17.6 | 25
  ART resumption: Lymphocytes/Leukocytes (low): number analyzed (Participants) | 17 | 8
  ART resumption: Lymphocytes/Leukocytes (low) | 11.8 | 0
  ART resumption: Monocytes/Leukocytes (high): number analyzed (Participants) | 17 | 8
  ART resumption: Monocytes/Leukocytes (high) | 64.7 | 50
  ART resumption: Monocytes (high) | 11.8 | 0
  ART resumption: Neutrophils (low): number analyzed (Participants) | 17 | 8
  ART resumption: Neutrophils (low) | 41.2 | 12.5
  ART resumption: Neutrophils/Leukocytes (high): number analyzed (Participants) | 17 | 8
  ART resumption: Neutrophils/Leukocytes (high) | 0 | 12.5
  ART resumption: Neutrophils/Leukocytes (low): number analyzed (Participants) | 17 | 8
  ART resumption: Neutrophils/Leukocytes (low) | 29.4 | 25
  Platelet count | 0 | 0

13. Primary Outcome: Percentage of Participants With Sustained Viremic Control (Human Immunodeficiency Virus [HIV] Ribonucleic Acid [RNA] Less Than [<]50 Copies Per Milliliter [Copies/mL]) During ATI Phase
Description: Percentage of participants with sustained viremic control (HIV RNA <50 copies/mL) during ATI phase were reported.
Time Frame: From Week 60 to Week 96
Population: The primary Efficacy Population (EP) included all participants who started antiretroviral (ARV) ATI at Week 60 and interrupted at least one dose of ART (Stage 2), regardless of the time or outcome of treatment interruption.
Measure: Number; unit: percentage of participants
Arm/Group | Ad26.Mos.HIV Vaccine or MVA Mosaic Vaccine | Placebo
Number analyzed (Participants) | 17 | 9
percentage of participants | 0 | 11.1

14. Primary Outcome: Duration of Sustained Viremic Control With HIV RNA <50 Copies/mL During ATI Phase
Description: Duration of sustained viremic control With HIV RNA <50 copies/mL during ATI Phase was reported.
Time Frame: From Week 60 to Week 96
Population: The primary EP included all participants who started ARV ATI at Week 60 and interrupted at least one dose of ART (Stage 2), regardless of the time or outcome of treatment interruption.
Measure: Mean (95% Confidence Interval); unit: weeks
Arm/Group | Ad26.Mos.HIV Vaccine or MVA Mosaic Vaccine | Placebo
Number analyzed (Participants) | 0 | 1
weeks |  | 27.7 [NA to NA] — Here NA refers that upper and lower limit of Confidence interval cannot be calculated for 1 participant.

15. Secondary Outcome: Total HIV Deoxyribonucleic Acid (DNA) Levels Over Time
Description: The total HIV DNA levels were assessed as a biomarker of the HIV reservoir.
Time Frame: From Week 60 to Week 96
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: copies/10E6 cells
Arm/Group | Ad26.Mos.HIV Vaccine or MVA Mosaic Vaccine | Placebo
Number analyzed (Participants) | 17 | 9
copies/10E6 cells
  Start of ATI | 34.83 (54.04) | 80.10 (117.36)
  6 Months post ATI | 47.24 (67.49) | 80.00 (72.52)

16. Secondary Outcome: Change in Cluster of Differentiation (CD)4 Count Over Time
Description: Change in CD4 count over time was reported. Assessment of residual HIV replication and viral reservoir in total CD4+ T cells was measured by quantitative real-time polymerase chain reaction (PCR).
Time Frame: Baseline and from Week 60 to Week 96
Population: The primary EP included all participants who started ARV ATI at Week 60 and interrupted at least one dose of ART (Stage 2), regardless of the time or outcome of treatment interruption. Here 'n' (number analyzed) signifies number of participants evaluable for specified categories.
Measure: Median (Inter-Quartile Range); unit: Median cells per cubic milliliters
Arm/Group | Ad26.Mos.HIV Vaccine or MVA Mosaic Vaccine | Placebo
Number analyzed (Participants) | 17 | 9
Median cells per cubic milliliters
  Baseline | 637 [545.0 to 757.0] | 531 [452.0 to 717.0]
  ATI | 602 [542.0 to 730.0] | 498 [465.0 to 545.0]
  ART: number analyzed (Participants) | 17 | 8
  ART | 661 [561.0 to 730.0] | 618 [485.0 to 775.5]
  Week 96 | 620 [556.0 to 753.0] | 538 [474.0 to 805.0]

17. Secondary Outcome: Time to Reinitiating ART
Description: Time to reinitiating ART was reported.
Time Frame: Up to Week 96
Population: The primary EP included all participants who started ARV ATI at Week 60 (Stage 2), regardless of the time or outcome of treatment interruption.
Measure: Mean (95% Confidence Interval); unit: Weeks
Arm/Group | Ad26.Mos.HIV Vaccine or MVA Mosaic Vaccine | Placebo
Number analyzed (Participants) | 17 | 9
Weeks | 5.4 [4.64 to 6.18] | 4.5 [3.14 to 5.93]

18. Secondary Outcome: Number of Participants With Acute Retroviral Syndrome Post-ARV ATI
Description: Number of participants with acute retroviral syndrome post-ARV ATI were reported.
Time Frame: From Week 60 to Week 96
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Ad26.Mos.HIV Vaccine or MVA Mosaic Vaccine | Placebo
Number analyzed (Participants) | 17 | 9
Participants | 0 | 0

19. Secondary Outcome: Duration of Acute Retroviral Syndrome Post-ARV ATI
Description: Duration of acute retroviral syndrome post-ARV ATI was reported.
Time Frame: From Week 60 to Week 96
Population: as for outcome 14
Measure: Median (Full Range); unit: weeks
Arm/Group | Ad26.Mos.HIV Vaccine or MVA Mosaic Vaccine | Placebo
Number analyzed (Participants) | 17 | 9
weeks | NA [NA to NA] — No acute retroviral syndrome was reported during the study. | NA [NA to NA] — No acute retroviral syndrome was reported during the study.

20. Secondary Outcome: Percentage of Participants With HIV Resistance to ARV Drugs Who Experienced Rebound Viremia After ARV ATI
Description: Percentage of participants with HIV resistance to ARV drugs who experienced rebound viremia after ARV ATI were reported. An HIV genotype test was done to evaluate and characterize HIV resistance to ARV drugs in participants who experience rebound viremia after ARV ATI.
Time Frame: From Week 60 to Week 96
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | Ad26.Mos.HIV Vaccine or MVA Mosaic Vaccine | Placebo
Number analyzed (Participants) | 17 | 9
percentage of participants | 35.3 | 22.2

21. Secondary Outcome: Percentage of Responders With Interferon-gamma (IFN-gamma) T Cell Responses Analyzed by Enzyme-linked Immunospot Assay (ELISpot) at Week 24, 26, 48, and 50
Description: Frozen peripheral blood mononuclear cell (PBMCs) was analyzed by interferon-gamma (IFN-gamma) (ELISpot). The response was defined as post-baseline value >P95 if baseline <P95 or missing or defined as post-baseline value >3-fold increase from baseline if baseline >=P95. The threshold for ELISpot test was based on the 95th percentile (P95) from the baseline values of participants on that test in the study.
Time Frame: At Week 24, 26, 48 and 50
Population: The Immunogenicity Population (IP) included all participants who were randomized and received at least 3 vaccinations according to the protocol-specified vaccination schedule, excluding the participant with a major protocol deviation. Here 'n' (number analyzed) signifies number of participants evaluable at specified time points.
Measure: Number; unit: percentage of responders
Arm/Group | Ad26.Mos.HIV Vaccine or MVA Mosaic Vaccine | Placebo
Number analyzed (Participants) | 17 | 9
percentage of responders
  HIV IFNg ENV pep pool (Clinical PTE): Week 24 | 70.6 | 11.1
  HIV IFNg ENV pep pool (Clinical PTE): Week 26 | 100 | 22.2
  HIV IFNg ENV pep pool (Clinical PTE): Week 48 | 70.6 | 22.2
  HIV IFNg ENV pep pool (Clinical PTE): Week 50: number analyzed (Participants) | 15 | 7
  HIV IFNg ENV pep pool (Clinical PTE): Week 50 | 80.0 | 0
  HIV IFNg ENV pep pool (Mos1): Week 26 | 94.1 | 0
  HIV IFNg ENV pep pool (Mos1): Week 50: number analyzed (Participants) | 15 | 7
  HIV IFNg ENV pep pool (Mos1): Week 50 | 100 | 0
  HIV IFNg ENV pep pool (Mos2): Week 26 | 58.8 | 0
  HIV IFNg ENV pep pool (Mos2): Week 50: number analyzed (Participants) | 15 | 7
  HIV IFNg ENV pep pool (Mos2): Week 50 | 66.7 | 0
  HIV IFNg ENV10 pep subpool (PTE): Week 26 | 11.8 | 0
  HIV IFNg ENV10 pep subpool (PTE): Week 50: number analyzed (Participants) | 15 | 7
  HIV IFNg ENV10 pep subpool (PTE): Week 50 | 20.0 | 0
  HIV IFNg ENV11 pep subpool (Mos1): Week 26 | 0 | 0
  HIV IFNg ENV11 pep subpool (Mos1): Week 50: number analyzed (Participants) | 15 | 7
  HIV IFNg ENV11 pep subpool (Mos1): Week 50 | 0 | 0
  HIV IFNg ENV11 pep subpool (Mos2): Week 26: number analyzed (Participants) | 14 | 7
  HIV IFNg ENV11 pep subpool (Mos2): Week 26 | 0 | 0
  HIV IFNg ENV11 pep subpool (Mos2): Week 50: number analyzed (Participants) | 15 | 7
  HIV IFNg ENV11 pep subpool (Mos2): Week 50 | 0 | 0
  HIV IFNg ENV11 pep subpool (PTE): Week 26 | 11.8 | 0
  HIV IFNg ENV11 pep subpool (PTE): Week 50: number analyzed (Participants) | 15 | 7
  HIV IFNg ENV11 pep subpool (PTE): Week 50 | 0 | 0
  HIV IFNg ENV12 pep subpool (Mos1): Week 26 | 5.9 | 0
  HIV IFNg ENV12 pep subpool (Mos1): Week 50: number analyzed (Participants) | 15 | 7
  HIV IFNg ENV12 pep subpool (Mos1): Week 50 | 0 | 0
  HIV IFNg ENV12 pep subpool (Mos2): Week 26: number analyzed (Participants) | 14 | 7
  HIV IFNg ENV12 pep subpool (Mos2): Week 26 | 0 | 0
  HIV IFNg ENV12 pep subpool (Mos2): Week 50: number analyzed (Participants) | 15 | 7
  HIV IFNg ENV12 pep subpool (Mos2): Week 50 | 0 | 0
  HIV IFNg ENV12 pep subpool (PTE): Week 26 | 11.8 | 0
  HIV IFNg ENV12 pep subpool (PTE): Week 50: number analyzed (Participants) | 15 | 7
  HIV IFNg ENV12 pep subpool (PTE): Week 50 | 6.7 | 0
  HIV IFNg ENV13 pep subpool (Mos1): Week 26 | 0 | 0
  HIV IFNg ENV13 pep subpool (Mos1): Week 50: number analyzed (Participants) | 15 | 7
  HIV IFNg ENV13 pep subpool (Mos1): Week 50 | 0 | 0
  HIV IFNg ENV13 pep subpool (Mos2): Week 26: number analyzed (Participants) | 14 | 7
  HIV IFNg ENV13 pep subpool (Mos2): Week 26 | 21.4 | 0
  HIV IFNg ENV13 pep subpool (Mos2): Week 50: number analyzed (Participants) | 15 | 7
  HIV IFNg ENV13 pep subpool (Mos2): Week 50 | 6.7 | 0
  HIV IFNg ENV13 pep subpool (PTE): Week 26 | 5.9 | 0
  HIV IFNg ENV13 pep subpool (PTE): Week 50: number analyzed (Participants) | 15 | 7
  HIV IFNg ENV13 pep subpool (PTE): Week 50 | 0 | 0
  HIV IFNg ENV14 pep subpool (Mos1): Week 26 | 17.6 | 0
  HIV IFNg ENV14 pep subpool (Mos1): Week 50: number analyzed (Participants) | 15 | 7
  HIV IFNg ENV14 pep subpool (Mos1): Week 50 | 20.0 | 0
  HIV IFNg ENV14 pep subpool (Mos2): Week 26: number analyzed (Participants) | 14 | 7
  HIV IFNg ENV14 pep subpool (Mos2): Week 26 | 14.3 | 0
  HIV IFNg ENV14 pep subpool (Mos2): Week 50: number analyzed (Participants) | 15 | 7
  HIV IFNg ENV14 pep subpool (Mos2): Week 50 | 6.7 | 0

22. Secondary Outcome: Percentage of Responders for Envelop (Env) Clade A, B, C and Mos1-specific Binding Antibody Titers
Description: The Env Clade A (92UG037), B (1990a), and C (Con C), (C97ZA.012) and Mos1- specific binding antibody titer were assessed using enzyme-linked immunosorbent assay (ELISA). The response was defined as post-baseline value greater than (>) lower limit of quantification (LLOQ) if baseline less than (<) LLOQ or missing or defined as post-baseline value >3-fold increase from baseline if baseline greater than or equal to (>=) LLOQ. The lower limits of quantification (LLOQs) for this assay were 625, 156.25, 625, 156.25 and 78.125 endotoxin units per milliliter (EU/mL) for Clade A (92UG037), Clade B (1990a), Clade C (Con C), Clade C (C97ZA.012) and Mos1 respectively.
Time Frame: At Week 24, 26, 48 and 50
Population: The IP included all participants who were randomized and received at least 3 vaccinations according to the protocol-specified vaccination schedule, excluding the participant with a major protocol deviation.
Measure: Number; unit: percentage of responders
Arm/Group | Ad26.Mos.HIV Vaccine or MVA Mosaic Vaccine | Placebo
Number analyzed (Participants) | 17 | 9
percentage of responders
  HIV ENV (gp140 T) A (92UG037.1) IgG-t Ab: Week 24 | 100 | 11.1
  HIV ENV (gp140 T) A (92UG037.1) IgG-t Ab: Week 26 | 100 | 0
  HIV ENV (gp140 T) A (92UG037.1) IgG-t Ab: Week 48 | 94.1 | 11.1
  HIV ENV (gp140 T) A (92UG037.1) IgG-t Ab: Week 50 | 100 | 0
  HIV ENV (gp140 T) B (1990a) IgG-t Ab: Week 24 | 100 | 0
  HIV ENV (gp140 T) B (1990a) IgG-t Ab: Week 26 | 100 | 0
  HIV ENV (gp140 T) B (1990a) IgG-t Ab: Week 48 | 100 | 0
  HIV ENV (gp140 T) B (1990a) IgG-t Ab: Week 50 | 100 | 0
  HIV ENV (gp140 T) C (ConC) IgG-t Ab: Week 24 | 94.1 | 0
  HIV ENV (gp140 T) C (ConC) IgG-t Ab: Week 26 | 70.6 | 0
  HIV ENV (gp140 T) C (ConC) IgG-t Ab: Week 48 | 82.4 | 0
  HIV ENV (gp140 T) C (ConC) IgG-t Ab: Week 50 | 94.1 | 0
  HIV ENV (gp140 T) C (ZA) IgG-t Ab: Week 4 | 76.5 | 0
  HIV ENV (gp140 T) C (ZA) IgG-t Ab: Week 16 | 82.4 | 0
  HIV ENV (gp140 T) C (ZA) IgG-t Ab: Week 24 | 82.4 | 0
  HIV ENV (gp140 T) C (ZA) IgG-t Ab: Week 26 | 82.4 | 0
  HIV ENV (gp140 T) C (ZA) IgG-t Ab; Week 48 | 64.7 | 0
  HIV ENV (gp140 T) C (ZA) IgG-t Ab: Week 50 | 76.5 | 0
  HIV ENV (gp140 T) Mos1 IgG-t Ab: Week 24 | 88.2 | 0
  HIV ENV (gp140 T) Mos1 IgG-t Ab; Week 26 | 100 | 0
  HIV ENV (gp140 T) Mos1 IgG-t Ab: Week 48 | 94.1 | 0
  HIV ENV (gp140 T) Mos1 IgG-t Ab: Week 50 | 94.1 | 0

23. Secondary Outcome: Percentage of Responders for Clade C (C97ZA.012) Env ELISA Immunoglobulin G1 (IgG1), IgG2, and IgG3 Glycoprotein (gp) 140 Binding Antibody
Description: Vaccine-induced binding antibody IgG1, IgG2, and IgG3 subclass responses were investigated using Clade C (C97ZA.012) specific ELISAs. The response was defined as post-baseline value >LLOQ if baseline <LLOQ or missing or defined as post-baseline value >3-fold increase from baseline if baseline >=LLOQ. The LLOQs for this assay were 12.3, 28.7, and 12.4, for IgG1, IgG2, and IgG3, respectively. Less participants were assessed for IgG2 responses due to lack of sample volume which led to a limit on the number of repeats that the analysis lab could perform. Reportable results were not generated for the remaining participants post vaccination.
Time Frame: Week 50
Population: The IP included all participants who were randomized and received at least 3 vaccinations according to the protocol-specified vaccination schedule, excluding the participant with a major protocol deviation. Here 'n' (number analyzed) signifies number of participants evaluable at specified time points.
Measure: Number; unit: percentage of responders
Arm/Group | Ad26.Mos.HIV Vaccine or MVA Mosaic Vaccine | Placebo
Number analyzed (Participants) | 17 | 9
percentage of responders
  HIV ENV (gp140 T) clade C (ZA) IgG-1 Ab: number analyzed (Participants) | 16 | 9
  HIV ENV (gp140 T) clade C (ZA) IgG-1 Ab | 68.8 | 0
  HIV ENV (gp140 T) clade C (ZA) IgG-2 Ab: number analyzed (Participants) | 3 | 0
  HIV ENV (gp140 T) clade C (ZA) IgG-2 Ab | 0 |
  HIV ENV (gp140 T) clade C (ZA) IgG-3 Ab: number analyzed (Participants) | 16 | 9
  HIV ENV (gp140 T) clade C (ZA) IgG-3 Ab | 18.8 | 11.1

24. Secondary Outcome: Breadth of T Cell Responses Analyzed by ELISPOT Assays
Description: Breadth of T cell responses was assessed at baseline (Week 0), Week 26, and Week 50 by ELISPOT assays.
Time Frame: Baseline (Week 0), Week 26 and 50
Population: as for outcome 22
Measure: Median (Full Range); unit: Median number of subpools
Arm/Group | Ad26.Mos.HIV Vaccine or MVA Mosaic Vaccine | Placebo
Number analyzed (Participants) | 17 | 9
Median number of subpools
  Baseline | 2.0 [0 to 7] | 3.5 [0 to 11]
  Week 26 | 10.0 [3 to 23] | 3.0 [0 to 8]
  Week 50 | 8.0 [4 to 12] | 3.0 [0 to 8]

25. Secondary Outcome: Percentage of Env Antibody-dependent Cellular Phagocytosis (ADCP) Glycoprotein (gp) Antibody Over Time
Description: The functionality of vaccine-induced antibody responses was investigated by the determination of ADCP. The response was defined as post-baseline value > limit of detection (LOD) if baseline <LOD or missing or defined as post-baseline value >3-fold increase from baseline if baseline >=LOD. The lower limits of detection (LODs) for this assay were 4.28 (phagocytic score) for Mos1.
Time Frame: At Week 24, 26, 48 and 50
Population: as for outcome 22
Measure: Median (Full Range); unit: percentage of ADCP gp antibody
Arm/Group | Ad26.Mos.HIV Vaccine or MVA Mosaic Vaccine | Placebo
Number analyzed (Participants) | 17 | 9
percentage of ADCP gp antibody
  Week 24 | 4.500 [0.00 to 37.60] | 0 [0.00 to 1.00]
  Week 26 | 18.200 [0 to 50.00] | 0 [0 to 0.80]
  Week 48 | 10.500 [0.0 to 44.20] | 0 [0 to 1.80]
  Week 50 | 20.500 [0 to 49.00] | 0 [0 to 12.90]

26. Secondary Outcome: Percentage of Responders for HIV Neutralizing Antibody (nAb)
Description: The functionality of vaccine-induced antibody responses was investigated by the determination of nAb activity in a virus neutralization assay (VNA) using TZM-bl cells and Env-pseudotyped viruses. The response was defined as post-baseline value >LLOQ.
Time Frame: Week 64
Population: as for outcome 22
Measure: Number; unit: percentage of responders
Arm/Group | Ad26.Mos.HIV Vaccine or MVA Mosaic Vaccine | Placebo
Number analyzed (Participants) | 17 | 9
percentage of responders | 100 | 0

ADVERSE EVENTS:
Time Frame: Up to Week 96
Description: FAS included all participants who were randomized and who received at least 1 dose of study vaccine or placebo.
Arm/Group | Ad26.Mos.HIV Vaccine or MVA Mosaic Vaccine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/17 | 0/9
Other Adverse Events (participants affected / at risk) | 15/17 | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ad26.Mos.HIV Vaccine or MVA Mosaic Vaccine (N=17) | Placebo (N=9)
Palpitations (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ad26.Mos.HIV Vaccine or MVA Mosaic Vaccine (N=17) | Placebo (N=9)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 1 | 0
Anogenital Dysplasia (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Feeling Hot (General disorders) | 3 | 0
Pyrexia (General disorders) | 1 | 2
Food Allergy (Immune system disorders) | 0 | 1
Anal Chlamydia Infection (Infections and infestations) | 1 | 0
Chlamydial Infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1
Oropharyngeal Gonococcal Infection (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Subcutaneous Abscess (Infections and infestations) | 0 | 1
Syphilis (Infections and infestations) | 1 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 4 | 1
Urethritis (Infections and infestations) | 0 | 1
Urethritis Chlamydial (Infections and infestations) | 0 | 1
Animal Bite (Injury, poisoning and procedural complications) | 1 | 0
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 1
Cd4 Lymphocytes Decreased (Investigations) | 1 | 0
Hepatic Enzyme Increased (Investigations) | 1 | 0
Liver Function Test Increased (Investigations) | 3 | 0
Weight Decreased (Investigations) | 1 | 0
Abnormal Loss of Weight (Metabolism and nutrition disorders) | 0 | 1
Folate Deficiency (Metabolism and nutrition disorders) | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Subgroup analyses were performed by Ad26 baseline seropositivity for the humoral (ie, binding antibody responses; Env ELISA IgG-t gp140) and cellular immune responses (ie, IFN T cell responses and epitope mapping), and by time to rebound (3 tertile subgroups) for both the humoral and cellular immune responses (all parameters). Due to the low number of participants in each subgroup, no firm conclusions could be made.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation.

DOCUMENTS (2):
  • Study Protocol (2017-10-11): https://cdn.clinicaltrials.gov/large-docs/06/NCT02919306/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-17): https://cdn.clinicaltrials.gov/large-docs/06/NCT02919306/SAP_001.pdf